CLINICAL TRIAL: NCT02246686
Title: A Randomised, Double-blind, Placebo-controlled Multi-centre Study to Investigate the Effectiveness and Safety of STW5-II as add-on Treatment for Induction of Remission in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Efficacy/Safety Pilot Study to Investigate Iberogast N's Efficacy in Mild to Moderate Colitis Ulcerosa Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17155; 2013-000891-13 (EudraCT Number)
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Colitis, Ulcerative
Keywords: Iberogast N; Mild to moderate ulcerative colitis; add-on therapy; efficacy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- STW5-II (Experimental): Half of study population, assigned randomly
  Interventions: Drug: STW5-II (Iberogast N, BAY98-7410)
- Placebo (Placebo Comparator): Half of study population, assigned randomly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STW5-II (Iberogast N, BAY98-7410) — Application over 12 weeks 20 drops three time daily
  Arms: STW5-II
Drug: Placebo — Application over 12 weeks 20 drops three time daily
  Arms: Placebo

SUMMARY:
The study will investigate efficacy of STW5-II as add-on therapy on the rate to remission in patients with mild to moderate ulcerative colitis in an acute flare.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate active ulcerative colitis (UC), i.e. Clinical Activity Index (CAI) ≥ 5 up to 10 points (including)
* Patients in whom the active UC is treated independent from any participation in the current study with oral mesalazine at least 14 days up to maximal 28 days before Visit 2
* Age between 18 to 80 years (including)
* UC may reach from left-sided colitis to pancolitis

Exclusion Criteria:

* Severe forms of UC (CAI > 10)
* Crohn's disease, infectious colitis or undetermined colitis
* Steroid dependence and steroid resistance
* Concomitant medication with oral steroids, oral or topic budesonide, biologicals, immune modifiers, immunosuppressants
* Antibiotics at screening visit, during the course of the study a short-term use in non-colitic afflictions is allowed, and is documented
* Prior medication with biologicals, immune modifiers and immunosuppressants < 3 month wash-out
* Total colectomy
* Known allergies to components of STW5-II
* Severe allergic diathesis
* Topical mesalazine application
* Known intolerance to azo dyes E110 and E151

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients being in remission at final visit | Week 12
  Responder definition for remission: Clinical Activity Index (CAI) ≤ 4
Change of endoscopic index (EI) | From baseline to week 12
Change of histological index (HI) based on Riley | From baseline to week 12
Proportion of patients reaching a clinical CAI ≤ 2 points | Week 12
Time to remission, defined as days from Day 0 until first remission is reached | Up to 12 weeks
  Responder definition for remission: Clinical Activity Index (CAI) ≤ 4
Time to sustained remission (CAI ≤ 2 points) defined as days from Day 0 until first sustained remission is reached | Up to 12 weeks
Number of patients who reached a remission at least once during the course of the study | Week 12
Number of patients who reached a sustained remission at least once during the course of the study | Week 12
Change from baseline of absolute CAI values to final visit | From baseline to week 12
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ-D) (German version) at final visit | From baseline to week 12
Change from baseline in Irritable Bowel Severity Score (IBSS) at final visit | From baseline to week 12
Change from baseline in EuroQol 5 dimensions questionnaire (EQ-5D) at final visit | From baseline to week 12
Mayo Score throughout the study | Up to 12 weeks
Change of of oral mesalazine dose throughout the study period | From baseline to week 12
Change in ulcerative colitis (UC) markers | From baseline to week 12
  Combination of four markers C-reactive protein (CRP), calprotectin, lactoferrin, polymorphonuclear (PMN) elastase for determination of parameters associated with acute flare of UC patients

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Germany (8):
  - Dachau, Bavaria
  - Hamburg, Hamburg
  - Lüneburg, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Lübeck, Schleswig-Holstein
  - Berlin
  - Essen